CLINICAL TRIAL: NCT00715572
Title: Combined Therapy With L-Thyroxine and L-Triiodothyronine Compared to L-Thyroxine Alone in the Treatment of Primary Hypothyroidism
Brief Title: Combined Therapy With L-Thyroxine and L-Triiodothyronine Compared to L-Thyroxine Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: The I.M. Sechenov Moscow Medical Academy, Department of Endocrinology, The I.M. Sechenov Moscow Medical Academy, Department of Endocrinology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: T3T42008; T3T42005
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Hypothyroidism
Keywords: hypothyroidism, treatment, thyroxine, triiodothyronine
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine; Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: thyroxine
- B (Active Comparator)
  Interventions: Drug: thyroxine and triiodothyronine

INTERVENTIONS:
Drug: thyroxine — monotherapy with thyroxine
  Arms: A
Drug: thyroxine and triiodothyronine — combination with thyroxine and triiodothyronine
  Arms: B

SUMMARY:
The objective of this study was to analyze the features of monotherapy with L-T4 in comparison with combined therapy with L-T4 and L-T3 in patients with primary hypothyroidism.

DETAILED DESCRIPTION:
We conducted a randomized controlled study with a crossover design in 36 premenopausal women with overt primary hypothyroidism (reduced T4 concentration accompanied by increased TSH concentration at the time of initial diagnosis) who did not receive thyroid hormones. All patients were divided into two groups: patients from Group A (n=20) were randomized to L-T4 in dose of 1,6 μg per kg, followed by combined L-T4 and L-T3; and 16 women from Group B received the combination of L-T4+L-T3 (the dose of L-T4 was reduced by 25 μg and replaced with 12,5 μg of L-T3), followed by monotherapy with L-T4. The treatment periods lasted for 6 months. Patients were examined at baseline and at the end of each treatment period.Blood samples were obtained to measure serum TSH, free T4, free T3, lipid profile, osteocalcin. Urine samples were collected to measure urinary deoxypyridinoline / creatinine ratio. 24-hour ECG-monitoring, osteodensitometry and psychological testing were also performed at baseline and at the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with overt primary hypothyroidism (reduced T4 concentration accompanied by increased TSH concentration at the time of initial diagnosis) who did not receive thyroid hormones

Exclusion Criteria:

* Peri- and postmenopause
* Pregnancy
* Major comorbidity
* Use of drugs that affect metabolism or bioavailability of thyroid hormones preparations.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2002-03; Primary Completion 2004-02 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
biochemical parameters | the end of each period of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Valentin V Fadeyev, Principal Investigator — Moscow Medical Academy, Department of Endocrinology